CLINICAL TRIAL: NCT03479060
Title: Continue or Stop Applying Wet Cupping (Al-Hijamah) in Migraine Headache: A Randomized Control Trial
Brief Title: Continue or Stop Applying Wet Cupping (Al-Hijamah) in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Assist.Prof. Department of Family Medicine, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBU-BAP-14/1-KA-057.
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Migraine Disorders; Migraine With Aura; Migraine Without Aura
Keywords: Wet cupping therapy; Migraine; MIDAS
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue WCT Application (Active Comparator): From the 3rd month to the 12th month Wet cupping applied as an intervention MIDAS was applied at the end of the 6th and 12th months.
  Interventions: Procedure: Wet Cupping
- Discontinue WCT Application (No Intervention): No intervention in this arm.Only MIDAS applied

INTERVENTIONS:
Procedure: Wet Cupping — cupping technique procedure was conducted in five phases:Primary suction,Area disinfection,Scarification,Bloodletting and secondary suction and Removing and dressing
  Arms: Continue WCT Application

SUMMARY:
This study evaluates the short and long-term effects of application of Wet Cupping Therapy (WCT) in the treatment of migraine headaches in adults.Half of the participants will continue WCT application and the other half will not.

DETAILED DESCRIPTION:
In literature, Cupping therapy(CT) has been shown to be used mostly for pain control and the majority of RCT studies have shown that CT has potential benefits in pain conditions. Previous studies have reported the effect of pain mediator substance-P, endorphins, encephalins and dynorphins on pain(1) In addition to pain control, it is recommended for use as additional treatment in neurological diseases such as paralysis, Parkinson's disease and stroke Studies have shown successful results in the short term with the application of CT for migraine and tension-type headaches (2,3) Methodology Study design and Patient selection Patients with a history of migraine diagnosis who presented at the Research Polyclinic of Karabuk University Training and Research Hospital for wet-cupping therapy in the period May 2016-January 2018 were included in the study. Patients were excluded if they had a history of head and neck surgery, a diagnosis of sinusitis, a diagnosis of fibromyalgia and inflammatory disease (rheumatism, infection etc.), were pregnant, had a diagnosis of cancer, bleeding disorder and widespread skin disease, malignant hypertension or any other disease which could cause headache. The diagnosis of migraine was confirmed by an experienced neurologist and the migraine type was determined. The medical treatments of the patients were reviewed and MIDAS was applied to determine the baseline score. In addition to the medical treatment, WCT was applied once a month, 3 times (Day 0, 30, 60). At the end of the 3rd month patients were allocated into two parallel arms. They were randomly assigned to the intervention group or control group in a double blind manner by the sealed opaque envelope technique. Intervention group continued WCT whereas patients in the control group discontinued the treatment. MIDAS was applied again at the end of the 6th and 12th months to both of the groups. Disability values in the 6th and 12th months were evaluated with MIDAS between those who continued treatment (Group 1) and those who did not (Group 2). Approval for the study was granted by Turgut Ozal University Ethics Committee, with number 99950669/236, dated 30.06.2014.Study design, application procedures and any possible side effects were explained to the study participants and informed consents obtained. All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

MIDAS The migraine disability score is a scale evaluating disability and loss associated with migraine. It consists of 7 questions, the 1st, 3rd and 5th of which evaluate the days lost from school, work, housework or leisure activities because of headaches in the last 3 months. The 2nd and 4th questions evaluate the number of additional days lost from work or housework in the last 3 months due to a reduction in productivity (defined as at least a 50% reduction in productivity). An additional two questions (MIDAS A and B) evaluate the frequency of headaches and the severity of the headaches using a visual analog scale (VAS), but these are not added to the total MIDAS score. The total MIDAS points are obtained from the total of the first 5 questions. Total points of 0-5 = 1st degree (very little or no restriction), 6-10 points =2nd degree (mild or occasional restriction), 11-20 points = 3rd degree (moderate level of restriction), and 21 + points = 4th degree (severe restriction).

ELIGIBILITY:
Creteria:Inclusion Criteria:

Subject has migraine headache

Exclusion Criteria:

History of head and neck surgery, Diagnosis of sinusitis Diagnosis of fibromyalgia and inflammatory disease (rheumatism, infection etc.) Diagnosis of cancer Diagnosis of bleeding disorder Malignant hypertension

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
MIDAS evaluation | At the end of the 12th month.
  Improvement in the Disability values which were evaluated with MIDAS

CONTACTS AND LOCATIONS:
Overall Officials: SULEYMAN ERSOY, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University Karabuk Research and Education hospital, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sajid MI. Hijama therapy (wet cupping) - its potential use to complement British healthcare in practice, understanding, evidence and regulation. Complement Ther Clin Pract. 2016 May;23:9-13. doi: 10.1016/j.ctcp.2016.01.003. Epub 2016 Feb 1. PMID 27157951
- [Background] Ahmadi A, Schwebel DC, Rezaei M. The efficacy of wet-cupping in the treatment of tension and migraine headache. Am J Chin Med. 2008;36(1):37-44. doi: 10.1142/S0192415X08005564. PMID 18306448
- [Background] Benli AR, Oruc MA. What is the difference of effectiveness of wet cupping therapy in migraine types?. Biomedical Research, 2017, 28.20.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03479060/SAP_001.pdf
  • Study Protocol (2017-03-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT03479060/Prot_002.pdf